CLINICAL TRIAL: NCT05191225
Title: Ultrafast Truxima Infusion in Non-Hodgkin's Lymphoma: Txagorapid Study - Intervention Pilot Study
Brief Title: Ultrafast Truxima Infusion in Non-Hodgkin's Lymphoma: Txagorapid Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laida Cuevas Palomares (Network)
Responsible Party: Sponsor-Investigator, Laida Cuevas Palomares, Dr. specialist in hematology and hemotherapy, Bioaraba Health Research Institute
Organization: Bioaraba Health Research Institute (Network)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TxagoRapid; 2019-001750-26 (EudraCT Number)
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: * Rapid infusion group After the administration of intravenous premedication (usually dexchlorpheniramine 5 mg IV and paracetamol 1 g IV), rituximab will be administered at standard dose (375 mg/m2 diluted in 250 ml of saline) administered in one hour, divided into: 10 first minutes at 450 mg/hour, and 50 minutes later at 720 mg/hour.
  * Ultrarapid infusion group After the administration of the premedication, the dose of rituximab will be administered at standard dose administered in half an hour, divided into: 10 first minutes at 450 mg/hour, and 20 minutes later at 1800mg/hour.
  * Ultrarapid plus infusion group After the administration of the premedication, the dose of rituximab will be administered at the standard dose administered in half an hour, divided into: 10 first minutes at 450 mg/hour, and 20 minutes later at 1800mg/hour.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rapid infusion group (Experimental): After the administration of intravenous premedication (usually dexchlorpheniramine 5 mg IV and paracetamol 1 g IV), rituximab will be administered at standard dose (375 mg/m2 diluted in 250 ml of saline) administered in one hour, divided into: 10 first minutes at 450 mg/hour, and 50 minutes later at 720 mg/hour.
  Interventions: Drug: RiTUXimab Injection [Truxima]
- Ultrarapid infusion group (Experimental): After the administration of intravenous premedication, the dose of rituximab will be administered at standard dose administered in half an hour, divided into: 10 first minutes at 450 mg/hour, and 20 minutes later at 1800mg/hour.
  Interventions: Drug: RiTUXimab Injection [Truxima]
- Ultrarapid plus infusion group (Experimental): After the administration of oral premedication, the dose of rituximab will be administered at the standard dose administered in half an hour, divided into: 10 first minutes at 450 mg/hour, and 20 minutes later at 1800mg/hour.
  Interventions: Drug: RiTUXimab Injection [Truxima]

INTERVENTIONS:
Drug: RiTUXimab Injection [Truxima] — 375 (mg/m2) / 60 minutes
  Arms: Rapid infusion group
Drug: RiTUXimab Injection [Truxima] — 375 (mg/m2) / 30 minutes
  Arms: Ultrarapid infusion group; Ultrarapid plus infusion group

SUMMARY:
The objective of this pilot study is therefore to assess the safety of Truxima ultrafast infusion within 30 minutes in patients with non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have tolerated the maximum rate of intravenous administration of rituximab (400 mg/h) in the first or second infusion.
* The last rituximab infusion must have occurred within the last 3 months.
* All patients receiving rituximab can be included, regardless of whether they receive rituximab as monotherapy or in combination with chemotherapy and regardless of the line in which they are receiving it.
* Patients will be included in both induction and maintenance treatment.
* All patients must sign the informed consent form.

Exclusion Criteria:

* Patients with initial absolute lymphocyte count >10x10^3 cells/µL.
* Patients who have presented hypersensitivity and severe adverse effects (grade II or higher) in the first or second infusion.
* Severe heart failure (NYHA class III-IV) or uncontrolled severe cardiac disease.
* Respiratory failure, severe uncontrolled COPD/asthma.
* Patients allergic to premedication: acetaminophen or polaramine.
* Severe active infection.
* Pregnant patients.
* Refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Infusional reactions | 24 hours
  Percentage of grade 2/3 or higher infusion reactions in rapid, ultrafast and ultrafast plus infusion compared to rituximab administration following standard clinical practice at standard rate of 400 mg/h.

CONTACTS AND LOCATIONS:
Overall Officials: Laida Cuevas Palomares, Principal Investigator — Bioaraba Health Research Institute
Locations (1):
- Hospital Universitario Araba- Sede Txagorritxu, Vitoria-Gasteiz, Alava, Spain